CLINICAL TRIAL: NCT02091713
Title: Musculoskeletal Injuries' Prediction Tool for Military Combatants in the Israeli Defense Force (FMS)
Brief Title: Musculoskeletal Injuries' Prediction Tool for Military Combatants in the Israeli Defense Force
Acronym: FMS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Oren Schwarz, Investigator in Heller institute of medical research, Sheba Medical Center
Other Study IDs: SHEBA-13-0529-BA-CTIL; 1294-2013 (Other: IDF)
Record Dates: First submitted 2014-03-12; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Cumulative Trauma Disorders
Keywords: FMS; functional movement screen
MeSH Terms: conditions — Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental/Functional movement screen: 300 subjects from three different combat units will undergo functional movement screening
  Interventions: Other: Functional movement screen

INTERVENTIONS:
Other: Functional movement screen — The subjects will undergo movement and balance screens, measures of power, demographic data and biopsychosocial measures. Injury data will be collected through physician exam, self-report, profile data, and healthcare utilization data. Injury data will be collected at baseline and for six iterations, every 60 days, over the course of one year following baseline. Based on the data collected, clinical prediction rules will be used to develop computerized algorithm to predict injury risk in these populations.

SUMMARY:
Emerging evidences indicate that performance on a variety of functional movement screens can identify athletes/soldiers at risk for injury. These field expedient tests have not been validated in a military setting or across different military occupational specialties. In this prospective study the investigators plan to screen 300 combatants for a 1-year time frame in order to validate the suggested algorithm of a list of modifiable and non-modifiable risk factors which are hypothesized to predict injury risk during the military service.

DETAILED DESCRIPTION:
Injury data will be collected through physician exam, self-report, profile data, and healthcare utilization data. Injury data will be collected at baseline and for six iterations, every 60 days, over the course of one year following baseline. Based on the data collected, clinical prediction rules will be used to develop computerized algorithm to predict injury risk in these populations. Moreover, these results will assist in creating individualized preventing physical training program.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-21 years old
* A combat medical profile according the IDF Medical Corp regulations
* Hebrew speaking and reading.

Exclusion Criteria:

* Currently seeking medical care for musculoskeletal injuries or has sought medical care for musculoskeletal injury in the last 30 days.
* Currently unable to participate in routine physical training due to injury in foot, ankle, knee, hip, neck, shoulder, elbow, wrist, or hand injury.
* Cardiac or pulmonary problems limiting physical activity.
* Known history of balance or visual impairment, neurological disorders, or chronic musculoskeletal conditions precluding their involvement in military training, physical training, or sports.
* Pregnancy, subjects that become pregnant during the course of the study will be excluded based on the different injury risk factors that are associated with musculoskeletal injury during pregnancy.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 300 soldiers in 3 units will be recruited and will undergo medical evaluation and functional movment screening as describes in the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Baseline surveillance | 1 week
  In this study all subjects will undergo a baseline assessment on recruitment, in which demographic, biopsychosocial, and physical data will be collected.
Injury surveillance | 1 year
  Yearly injury surveillance will be conducted on a 2-month basis in which the research team will prospectively collect data on any injury occurrence and medical health utilization among the study's subjects.

SECONDARY OUTCOMES:
Physical assessment | 1 year
  The physical assessment of risk factors will include the following 8 tests: foot structure and mobility (foot length, seated and standing AHI), assessment of functional movement (FMS), lower extremity power (SLVJ), hop testing, lower quarter Y-Balance Test (LQYBT), and upper quarter Y Balance test (UQYBT), ankle dorsiflexion, and the 240m shuttle run as detailed.
Demographic and biopsychosocial data | 1 week
  Demographic and biopsychosocial data collection will include general information, such as: age, gender, anthropometrics (height, weight), past medical history previous sport engagements, injury in the last 12 months, past physical activities and levels, smoking status, marital status, and educational level. In addition to these demographic variables all subjects will answer questions related to biopsychosocial factors associated with injury.
  This includes questions related to job/life satisfaction, numeric pain ratings associated with depression, anxiety, frustration, anger, and fear, and completion of the patient health questionnaire (PHQ-9) which will help in determining the influence of indicators of depression on future injury risk.

CONTACTS AND LOCATIONS:
Overall Officials: Oren Schwarz, M.D, Principal Investigator — Heller institute of medical research
Locations (1):
- Heller institute of medical research, Tel Litwinsky, Israel